CLINICAL TRIAL: NCT04659395
Title: How to Develop a Training Program for Nurses in Ultrasound Guided Femoral - a Methodology Study
Brief Title: How to Develop a Training Program for Nurses in Ultrasound Guided Femoral Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: University of South-Eastern Norway (Other)
Responsible Party: Principal Investigator, Espen Lindholm, Consultant, Sykehuset i Vestfold HF
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 533039
Record Dates: First submitted 2020-11-12; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Hip Fractures; Ultrasound Therapy; Complications; Pain, Acute
Keywords: Task shifting; Ultrasound guided; Training; Education; Emergency department; Registered nurse; Nerve block; Hip fracture
MeSH Terms: conditions — Hip Fractures; Acute Pain; Emergencies

STUDY DESIGN:
Intervention Model Description: A methodology study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emergency nurses (Other): Emergency nurses who are trained in an one-day course
  Interventions: Other: Emergency nurses

INTERVENTIONS:
Other: Emergency nurses — Emergency nurses who are trained for one-day in ultrasound-guided femoral nerve block

SUMMARY:
In this study the intervention consists of a one-day-training program for nurses and three supervised ultrasound guided femoral nerve block (UGFNB) per registered nurse.

The training consists of an instruction movie, one-day on-site-simulation and practical examination. The nurses are watching an instruction video and review current local guidelines for UGFNB in advance. The one-day training is situated in a simulation center and consists of theoretical and practical training divided into; infection prevention, anatomy, use of ultrasound and prevention and treatment of complications. A ultrasound model (Gen II Femoral Vascular Access and Regional Anesthesia Ultrasound Training Model) and a living human model is used to examine the femoral nerve and the neighboring structures using ultrasound. At the end of the one-day course, the nurses attends a practical examination with the researchers and anesthesiologists observing, to assure that they could perform the UGFNB procedure correctly. To pass the exam and be able to move on to the supervised blocks in real patients, there has to be a consensus between the researchers and anesthesiologist that they had sufficient knowledge and practical skills. 1) Sterile procedure 2) Management of the ultrasound machine and oral description of the anatomic surroundings in the groin area 3) Preparation of the local anesthetics and performance of an UGFNB. They also have to do an oral presentation in how they would perform a cardiopulmonary resuscitation procedure and how to manage complications / toxic reactions. Approved exam required at least seven points. This study will explore if a one-day course as described above is adequate, sufficient and maintains the safety framework of performing UGFNB in nurses

DETAILED DESCRIPTION:
Acute pain is a common reason for patients admitted to Emergency Departments (ED) . Globally over 1 million hip fractures occur yearly , a trauma that is close related with acute distinct pain in the proximal part of the affected extremity. Experiencing severe pain is associated with increased length of stay, higher risk of delirium, movement restriction, difficulties with mobilization and reduced health related quality of life. There is considerable research regarding patients' satisfaction with their ED experiences. These studies indicate that patient dissatisfaction with the stay at ED has been an international challenge over several years . Disapproval such as; pain management , but also limited information on potential latency before further treatment and poor explanation about the causes and treatment of the condition is prominent.

Pain control can be difficult , and often requires advanced nursing and physician care due to co-morbidity . Inadequate analgesia appear to be risk factors for delirium in frail older adults, and research indicates that total avoiding opioids or using very low or high doses of opioids may increase the risk of delirium. Therefore, optimizing acute pain management is important. Ultrasound Guided Femoral Nerve block (UGFNB) performed in hip fracture patients is a valuable alternative to systemic analgesic, as it provides analgesia to the fractured area, thereby facilitating reduction in opioid administration. Traditionally, an UGFNB is performed by an anesthesiologist. Recently, several examples of task shifting from physicians to nurses are described with no significant difference in successful treatment results with equal patients satisfaction and safety as physician performed procedures. Task shifting approach is endorsed by the World Health Organization (WHO) in order to make more efficient use of the available human resource of health. A recent report from the European Union (EU) states that implementation of task shifting has been rarely evaluated and limited documented. Therefore, we need studies to examine the methodology in how we can train nurses in the ED to take more responsibility for assessing and treating patients.

In the study we aime to;

1. describe a methodology for a training course for nurse led UGFNB.
2. evaluate if the training process resulted in a safe and successful UGFNB.

Data which will be collected are

1. ASA classification (ASA Physical Status Classification System )
2. Length of stay
3. Morbidity

   * Hospital acquired pneumonia
   * Acute myocardial infarction (AMI)
   * Acute renal failure
   * Respiratory failure
4. Complication rate, number of;

   * intravasal injection - visually + circulatory and neurological symptoms
   * hematoma - defined as a new tumor > 2 cm in the groin / injection site measured by ultrasound
   * Neurologic systemic outcomes / symptoms / paresthesia that have occurred after admission and which persist until discharge.
   * Allergic reaction
5. Number of total morphine equivalents, mg (iv/po) administered prehospital and during Emergency Department stay
6. Patients physical characteristic (physical examination; gender, age, height, weight, , blood pressure, heart rate, SpO2 (oxygen saturation) and use of oxygen will be noted together with current disease

A short, but personal interview with the patients having received an UGFNB by a study nurse can describe both the service received and the patient's experience with it. The interviews will be performed after the patient has been relieved of pain. The PhD (Philosophiae Doctor)-candidate, not the study nurse having performed the nerve block, will conduct the interviews. The patients will be asked whether the nerve block relieved them of pain, how they experienced the procedure and the fact that it was performed by a nurse had any relevance. Also, the PhD-candidate will interview the patient at a later point during the hospital stay for a second time to compare the answers

The study nurses and the anesthesiologists that has supervised the nurses will be presented with a questionnaire after each UGFNB conducted. The PhD-candidate will hand out the questionnaire immediately after the FNB is conducted by a study nurse. The items in the questionnaire include feasibility and success of the procedure and are identical for nurses and anesthesiologists.

Finally, each study nurse will do three UGFNB with supervision by an anesthesiologist before we start inclusion in a later randomized controlled trial. Five study nurses will be included and fifteen patients.

The inclusion criteria for patients will be:

* Patients arriving at the ED diagnosed with a hip fracture (radiological confirmed)
* ASA- classification 1-4
* Written and verbal informed consent by patient

Exclusion criteria for patients will be:

* Patients with; dementia, without ability to give informed consent and other cognitively challenges needed to participate in this study (at the discretion of the study nurse)
* Known allergies to local anesthetic (Ropivacaine) used in UGFNB
* Use of anticoagulants or platelet inhibitors. Acetylsalicylic acid and dipyridamole is allowed. If a recent (last 2 hours) INR( international normalized ratio) is below <1.5 the patient can be included.
* Pregnant
* Age <18 years
* Severe head injury which leads to significant loss of consciousness (GCS <12)
* >10 mg or more morphine administrated pre-hospital
* Skin lesions/infection at presumed block site
* Patients admitted with other suspected or verified fractures, except small fractures in hands and foots.

Verbal and written informed consent The study nurses will inform the patients by oral and written information and inclusion and intervention of the patient will start after written consent.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses or registered nurses with continuing education in acute nursing or geriatrics
* The nurses need to be aware that it will increase the workload in beginning of the project.
* Registered nurse has to be senior staff experienced i.e. worked in the ED
* Motivated to take on a new task in the ED
* Certificated in advanced CPR
* Familiar with routines in the ED and the relevant patient group
* They must be willing to be a part of this project for approximately 12 months.
* Working at least 75%.

Exclusion Criteria:

* Refuse to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Cumulative Numerical Rating Scale (NRS) - during passive movement at 120 minutes after start of procedure, measured by 5 timepoints | 120 minutes
  Cumulative Numerical Rating Scale (NRS) - during passive movement (30 degree flexion in the fractured hip) in patients with hip fracture during stay in the ED at 120 minutes after admission, measured by five time Points; At the end of procedure, 30 min.-, 60 min.-, 90 min.- and 120 min after start of procedure. NRS score: 0 is no pain and 10 is the worst pain.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) - during passive movement at baseline | At baseline (timepoint 0)
  Numerical Rating Scale (NRS) - during passive movement (30 degree flexion in the fractured hip) in patients with hip fracture during stay in the ED at baseline (inclution of patient) NRS score: 0 is no pain and 10 is the worst pain.
Numerical Rating Scale (NRS) - during passive movement after 30 minutes | After 30 minutes from baseline
  Numerical Rating Scale (NRS) - during passive movement (30 degree flexion in the fractured hip) in patients with hip fracture during stay in the ED after 30 minutes from baseline NRS score: 0 is no pain and 10 is the worst pain.
Numerical Rating Scale (NRS) - during passive movement after 60 minutes | After 60 minutes from baseline
  Numerical Rating Scale (NRS) - during passive movement (30 degree flexion in the fractured hip) in patients with hip fracture during stay in the ED after 60 minutes from baseline NRS score: 0 is no pain and 10 is the worst pain.
Numerical Rating Scale (NRS) - during passive movement after 90 minutes | After 90 minutes from baseline
  Numerical Rating Scale (NRS) - during passive movement (30 degree flexion in the fractured hip) in patients with hip fracture during stay in the ED after 90 minutes from baseline NRS score: 0 is no pain and 10 is the worst pain.
Numerical Rating Scale (NRS) - during passive movement after 120 minutes | After 120 minutes from baseline
  Numerical Rating Scale (NRS) - during passive movement (30 degree flexion in the fractured hip) in patients with hip fracture during stay in the ED after 120 minutes from baseline NRS score: 0 is no pain and 10 is the worst pain.
Hematoma | 24 hours
  Hematoma - defined as a new tumor > 2 centimeter in the groin / injection site measured by ultrasound, Yes or no
Intravasal injection | 24 hours
  Intravasal injection - visually + circulatory and neurological symptoms, yes or no
Patient experience- description of pain | 24 hours
  Patient experience of pain- During rest and motion measured by a 1-5 scale
Patient satisfaction- waiting time to pain relief | 24 hours
  Patiens experiences on waiting time to pain relief measured in a scale form 1-5
Patient satisfaction- information | 24 hours
  Patient experiences on information measured in a scale form 1-5
Patient satisfaction- description of pain before the procedure | 24 hours
  Patient experience on pre-procedure pain measured by 1-5 scale
Patient satisfaction- description of pain after the procedure | 24 hours
  Patient satisfaction- description of pain after the procedure measured by 1-5 scale
Patient satisfaction- safety | 24 hours
  Patient satisfaction- description of patient reported feeling of safety during nurse led procedure measured by a 1-5 scale
Patient satisfaction-effect of procedure | 24 hours
  Patient satisfaction regarding reduction of pain after the procedure measured by a 1-5 scale
Patient satisfaction-hearing status | 24 hours
  Patient satisfaction hearing status measured by a 1-4 scale
Self reported-registered nurse- complexity | approximately 2 hours
  Complexity of procedure measured by scale 1-5
Self reported-registered nurse-success | approximately 2 hours
  Success of procedure measured by 1-5 scale
Self reported-registered nurse-Recognition of anatomic structures | approximately 2 hours
  Recognition of anatomic structures at ultrasound, measured by a 1-4
Self reported-registred nurse-spread of anesthesia | approximately 2 hours
  Spread of anesthesia, measured by a 1-4 scale
Self reported-registered nurse- patient benefit from procedure | approximately 2 hours
  Patient benefit of procedure measured by a 1-5 scale
Self reported-Anesthesiologist-complexity | approximately 2 hours
  Complexity of procedure measured by scale 1-5
Self reported-Anesthesiologist-success | approximately 2 hours
  Success of procedure measured by a 1-5 scale
Self reported-Anesthesiologist-Recognition of anatomic structures | approximately 2 hours
  Recognition of anatomic structures at ultrasound measured by a 1-4 scale
Self reported-Anesthesiologist-spread of anesthesia | approximately 2 hours
  Spread of anesthesia, measured by a 1-4 scale
Self reported-Anesthesiologist-Patient benefit of procedure | approxemitely 2 hours
  Patient benefit of procedure measured by a 1-5 scale

CONTACTS AND LOCATIONS:
Overall Officials: Elin saga, Nurse, Principal Investigator — The Hospital of Vestfold
Locations (1):
- Vestfold Hospital Trust, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No
No plan for sharing IPD

REFERENCES:
- [Background] Dochez E, van Geffen GJ, Bruhn J, Hoogerwerf N, van de Pas H, Scheffer G. Prehospital administered fascia iliaca compartment block by emergency medical service nurses, a feasibility study. Scand J Trauma Resusc Emerg Med. 2014 Jun 23;22:38. doi: 10.1186/1757-7241-22-38. PMID 24957807
- [Background] Mandy, L. . Nurse-led femoral nerve service for patients with fractured neck of femur. Advanced Nursing Practice in Pain Management. C. E. e. al., John wiley and sons: (2009)16.
- [Background] Ketelaars R, Stollman JT, van Eeten E, Eikendal T, Bruhn J, van Geffen GJ. Emergency physician-performed ultrasound-guided nerve blocks in proximal femoral fractures provide safe and effective pain relief: a prospective observational study in The Netherlands. Int J Emerg Med. 2018 Mar 2;11(1):12. doi: 10.1186/s12245-018-0173-z. PMID 29500558
- [Background] Layzell M. Nurse-led femoral nerve block service for patients with fractured neck of femur. 2010 05.02.18. In: Advancing nursing practice in pain management [Internet]. Chichester, West Sussex; Ames, Iowa: Blackwell Pub.; [16]
- [Background] WHO (2008). Task Shifting - Global Recommendations and Guidelines. WHO. Geneva, Switzerland., WHO Document Production Services: 96.